CLINICAL TRIAL: NCT01306669
Title: Vaccination of HIV-uninfected Pregnant Women With Trivalent Influenza Vaccine in the Prevention of Influenza Illness During Early Infancy and in Mothers: Randomized Controlled Phase III Trial Evaluating Safety, Immunogenicity and Efficacy
Brief Title: Influenza Vaccine Trial in HIV Uninfected Pregnant Women
Acronym: MatfluHIVneg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Emory University (Other); University of Colorado, Denver (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Shabir Madhi, Medical officer, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Maternal_flu_HIVneg_101106
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent influenza vaccine (Active Comparator): Single dose administration of trivalent influenza vaccine prior to onset of influenza season
  Interventions: Biological: Trivalent influenza vaccine
- Normal saline (Placebo Comparator)
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Trivalent influenza vaccine — single dose of 0.5ml of Trivalent influenza vaccine for season will be administered into deltoid muscle of non-dominant arm
  Other Names: Vaxigrip
  Arms: Trivalent influenza vaccine
Biological: Normal saline — Single dose of 0.5ml of normal saline will be administered into deltoid muscle of non-dominant arm
  Other Names: NaCl
  Arms: Normal saline

SUMMARY:
Randomised, double blind, placebo controlled trial to assess safety, immunogenicity and efficacy of Trivalent Influenza vaccine in HIV uninfected pregnant women

DETAILED DESCRIPTION:
Acute respiratory illness is a significant contributor to neonatal mortality and the leading cause of under- 5 childhood mortality particularly during infancy. Infants under 6 months of age have the highest rate of excess influenza-associated hospitalization in industrialized countries among paediatric age groups. Determining the contribution of influenza to early childhood morbidity and mortality in sub-Saharan Africa and the potential to prevent influenza disease through vaccination may contribute to reducing childhood deaths; since influenza illness is a vaccine preventable disease for which vaccines are developed, licensed and available at reasonable cost. Unfortunately, infants at highest risk for serious disease are those under 6 months of age, for whom trivalent inactivated influenza vaccine (TIV) is poorly immunogenic and not licensed. As pregnant women also have an increased risk of serious illness (3.3-5.5 fold for hospitalization for influenza-associated acute cardio-respiratory illness) from influenza infection, one strategy to prevent the complications of influenza in pregnant women and young infants is through maternal TIV immunization, which is recommended by the WHO. This could result in direct protection of the women and protection of the young infant consequent to transplacental transfer of TIV induced antibody.

Barriers to administration of vaccines during pregnancy including lack of information on effectiveness and concerns about safety probably explain the virtual non-existent use of TIV in pregnant women from low-middle income countries. Recently data have become available from Bangladesh in which the benefit of maternal TIV vaccination was demonstrated by a 63% (95%CI 5 to 85) reduction in laboratory-confirmed influenza illness in infants under 24 weeks of age in children born to mothers vaccinated with TIV and a 36% reduction in clinical illness in vaccinated mothers.

Much of the influenza virus-associated morbidity and mortality may be due to the synergistic lethality of influenza with bacterial pathogens leading to pneumonia as well as other viral co-infections. Superimposed bacterial infections, especially Streptococcus pneumoniae, contribute to a large proportion of pneumonia deaths associated with influenza illness during pandemics.

The overall aim of this project is to evaluate the safety, immunogenicity and efficacy of TIV vaccination of HIV-uninfected pregnant women in preventing influenza related illness in their young infants, as well as among the women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years to less than 39 years.
* Gestational age greater than or equal to 20 weeks to less than 34 weeks documented by the approximate date of the last menstrual period and corroborated by physical exam.
* Documented to be HIV-1 uninfected on two assays used in the PMTCT program undertaken within 12 weeks of study enrolment.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of study.

Exclusion Criteria:

* Receipt of TIV, other than through the study, during the current influenza season documented by medical history or record.
* Receipt of any live licensed vaccine less than or equal to 28 days or inactivated licensed vaccine (except for tetanus toxoid vaccine) less than to equal to 14 days prior to study-vaccine.
* Participants in the nested immunogenicity cohort cannot receive ANY vaccine (including tetanus toxoid) within 14 days of the study-vaccine.
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) less than or equal to 28 days prior to vaccination in this study, or expects to receive another non-licensed agent before delivery unless study approval is obtained.
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 38 degrees C ≤ 24 hours prior to study entry.
* Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or has immunosuppression as a result of an underlying illness or treatment.
* Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤ 12 weeks of study entry, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) ≤ 12 weeks before study entry (nasal and topical steroids are allowed).
* Receipt of corticosteroids for preterm labor ≤ 14 days before study entry.
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.
* Receipt of IL2, IFN, GMCSF or other immune mediators ≤ 12 weeks before enrollment.
* Uncontrolled major psychiatric disorder.
* History of a severe adverse reaction to previous TIV.
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Pregnancy complications (in the current pregnancy) such as pre-term labor, hypertension (systolic blood pressure ≥ 140 and/or diastolic blood pressure ≥ 90 mm Hg) and pre-eclampsia.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2116 (Actual)
Dates: Start 2011-03-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The number of laboratory-confirmed influenza cases in infants born to mothers who received TIV or placebo will be used to determine efficacy of TIV vaccination of pregnant women against laboratory-confirmed influenza illness in their infants | 24 weeks of age
  All infants (up to 24 weeks of age) born to women enrolled on trial will be assessed by study staff if they have any signs or symptoms (including fever, hospitalisation, apnea, cough, nasal catarrh/ congenstion, tachypnea) which could indicate influenza like illness. Nasopharyngeal aspirate samples collected at illness visits will be processed for viruses using real time reverse transcriptase-polymerase chain reaction (rRTPCR) assays.
Humoral and cell-mediated immune (CMI) responses to influenza strains in the vaccine will be measured to assess the immunogenicity of TIV in pregnant women vaccinated between 20-34 weeks of gestational age | one month post vaccination, delivery (+7 days), 24 weeks post natal
  Humoral immunity will be measured by hemagglutination inhibition (HAI) assay. Blood will be collected at enrolment (pre-vaccination), one month post vaccination, delivery (+7 days) and 24 weeks post delivery. Humoral immune response definitions: HAI titers < 1:10 = seronegative; ≥ 1:10 = seropositive; > 1:40 = protected against influenza; Response to TIV = serconversion (from <1:10 to ≥1:10) and/or 4-fold increase of HAI titers. Cell mediated immunity will be measured by ELISPOT response to TIV. Blood will be collected at enrollment (pre-vaccination) and one month post vaccination.

SECONDARY OUTCOMES:
Hemagglutinin (HA) antibody measurements in blood taken from mother and infants up to 24 weeks post delivery will be used to assess kinetics of transplacentally acquired antibodies | Birth (+7 days), 8, 16 & 24 weeks of age
  Hemagglutinin (HA) antibody measurements in blood taken from mother at birth and infants at birth, 8,16 and 24 weeks post delivery will be used to assess kinetics of transplacentally acquired antibodies
Clinical influenza like illnesses in infants born to TIV and placebo recipients will be used to assess efficacy of TIV in pregnant women against ILI in their infants | 24 weeks of age
  All infants participants will have illness visits conducted if they have any signs or symptoms which may be suggestive of influenza-like illness (ILI). Infants with ILI, but with no Influenza virus isolated from nasopharyngeal aspirates will be classified as having clinical ILI. Clinical ILI cases in infants of TIV and placebo recipients will be compared to determine efficacy of TIV against ILI.
The number of laboratory-confirmed influenza illnesses in maternal participants during pregnancy and for 24 weeks post-partum will be used to assess efficacy of TIV against laboratory confirmed influenza | 24 weeks post delivery
  All maternal participants with signs and/ or symptoms of influenza like illness (ILI) will have nasopharyngeal and oropharyngeal swabs collected at illness visits and processed by rRTPCR assays. Participants from whom influenza virus is isolated at illness visits will be included in analysis to evaluate the efficacy of TIV against laboratory-confirmed influenza illness in mothers during pregnancy and until 24 weeks post-partum
The number of maternal participants who have ILI in whom influenza is not isolated from NP or OP swabs will be used to determine efficacy of TIV against clinical ILI in mothers | 24 weeks post delivery
  Maternal participants will be followed up from enrollment until 24 weeks post delivery for any influenza like illness. Women who have ILI episodes during which influenza is not isolated from NP/ OP swabs will be included in analysis to define the efficacy of TIV against protocol defined clinical ILI in women during pregnancy and until 24 weeks post-partum
Infants born to TIV/ placebo recipients will have nasopharyngeal swabs collected at 8, 16 and 24 weeks of age to determine acquisition of pneumococcal carriage | 24 weeks of age
  Infants born to women on immunogenicity cohorts will have nasopharyngeal swabs collected at 8, 16 and 24 weeks of age. The swabs will be processed for pneumococcal carriage and results will be used to define the efficacy of TIV against acquisition of pneumococcal carriage in infants up to 24 weeks of chronological age

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Study Chair — University of Witwatersrand, South Africa; Keith P Klugman, MD, PhD, Study Director — Emory University; Adriana Weinberg, Study Director — University of Denver
Locations (1):
- RMPRU, Chris Hani Baragwanath Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Motsoeneng BM, Dhar N, Nunes MC, Krammer F, Madhi SA, Moore PL, Richardson SI. Hemagglutinin Stalk-Specific Fc-Mediated Functions Are Associated With Protection Against Influenza Illness After Seasonal Influenza Vaccination. J Infect Dis. 2024 Dec 16;230(6):1329-1336. doi: 10.1093/infdis/jiae241. PMID 38743692
- [Derived] Amin AB, Nunes MC, Tapia MD, Madhi SA, Cutland CL, Wairagkar N, Omer SB; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Immunogenicity of influenza vaccines administered to pregnant women in randomized clinical trials in Mali and South Africa. Vaccine. 2020 Sep 22;38(41):6478-6483. doi: 10.1016/j.vaccine.2020.07.020. Epub 2020 Aug 29. PMID 32868130
- [Derived] Madhi SA, Cutland CL, Downs S, Jones S, van Niekerk N, Simoes EAF, Nunes MC. Burden of Respiratory Syncytial Virus Infection in South African Human Immunodeficiency Virus (HIV)-Infected and HIV-Uninfected Pregnant and Postpartum Women: A Longitudinal Cohort Study. Clin Infect Dis. 2018 May 17;66(11):1658-1665. doi: 10.1093/cid/cix1088. PMID 29253090
- [Derived] Nunes MC, Cutland CL, Jones S, Downs S, Weinberg A, Ortiz JR, Neuzil KM, Simoes EAF, Klugman KP, Madhi SA. Efficacy of Maternal Influenza Vaccination Against All-Cause Lower Respiratory Tract Infection Hospitalizations in Young Infants: Results From a Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1066-1071. doi: 10.1093/cid/cix497. PMID 28575286
- [Derived] Madhi SA, Nunes MC, Weinberg A, Kuwanda L, Hugo A, Jones S, van Niekerk N, Ortiz JR, Neuzil KM, Klugman KP, Simoes EAF, Cutland CL; Maternal Flu Trial (Matflu) Team. Contribution of Serologic Assays in the Evaluation of Influenza Virus Infection Rates and Vaccine Efficacy in Pregnant Women: Report From Randomized Controlled Trials. Clin Infect Dis. 2017 Jun 15;64(12):1773-1779. doi: 10.1093/cid/cix241. PMID 28369198
- [Derived] Nunes MC, Cutland CL, Jones S, Hugo A, Madimabe R, Simoes EA, Weinberg A, Madhi SA; Maternal Flu Trial Team. Duration of Infant Protection Against Influenza Illness Conferred by Maternal Immunization: Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2016 Sep 1;170(9):840-7. doi: 10.1001/jamapediatrics.2016.0921. PMID 27380464
- [Derived] Madhi SA, Cutland CL, Kuwanda L, Weinberg A, Hugo A, Jones S, Adrian PV, van Niekerk N, Treurnicht F, Ortiz JR, Venter M, Violari A, Neuzil KM, Simoes EA, Klugman KP, Nunes MC; Maternal Flu Trial (Matflu) Team. Influenza vaccination of pregnant women and protection of their infants. N Engl J Med. 2014 Sep 4;371(10):918-31. doi: 10.1056/NEJMoa1401480. PMID 25184864